CLINICAL TRIAL: NCT03666559
Title: Treatment With Azacitidine of Recurrent Gliomas With IDH1/2 Mutation
Acronym: AGIR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140910J; 2016-002822-35 (EudraCT Number)
Record Dates: First submitted 2018-06-15; First posted 2018-09-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Recurrent IDH1/2 Mutated Glioma
Keywords: Glioma; IDH1/2; Azacitidine; PFS
MeSH Terms: conditions — Glioma | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine (Experimental): Azacitidine is administered by sub-cutaneous injection at 75 mg/m2 per day for seven consecutive days every 4 weeks until progression, intolerance or end of the study.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Chemotherapy
  Other Names: Vidaza

SUMMARY:
Glioma are the most commun frequent brain tumour. Mutation of Isocitrate DeHydrogenase IDH1 or IDH2 genes affect 40% of gliomas, mostly grade II and III gliomas. Despite IDH mutated gliomas (IDHm glioma) have a better prognosis compared to the IDH wild type counterparts, they invariably recur after standard treatment with radiotherapy and alkylating agent. IDH mutation results in the accumulation of D-2 hydroxyglutarate (D2HG) produced by the IDH mutant enzyme. D2HG acts as a competitive inhibitor of the alphaketoglutarate cofactor in a wide range of cellular reactions, including Ten-eleven translocation (TET) family enzymes and histone demethylases, resulting in DNA hypermethylation (CIMP phenotype) and histone hypermethylation. Preclinical data have shown a dramatic anti-tumor effect of hypomethylating drugs as 5-azacytidine on IDH1 mutated human gliomas. These hypomethylating drugs are routinely used in myelodysplasic syndrome (MDS) and are well tolerated.

The AGIR Trial will be a phase II, non-comparative, open label, non randomised monocentric trial evaluating efficacy of a treatment by azacitidine in recurrent IDHm gliomas. The main objective is to evaluate the efficacy of azacitidine according to the RANO criteria on progression-free survival at 6 months, evaluated according to the RANO criteria. Given the slow mode of action of treatment, it is proposed to include only patients whose life expectancy at inclusion is greater than 9 months.

A 6-month progression-free survival of less than 15% will be inefficient. The minimum efficiency must be at least 30%. An interim analysis (according to Fleming's method) will be performed when 19 patients have been included and followed up to 6 months. If the interim analysis is inconclusive, 36 additional patients will be included. The maximum number of analysable patients to include is 55.

DETAILED DESCRIPTION:
Scientific justification:

Gliomas are the most frequent brain tumors. Prognosis is poor. It depends on the histological grade (I to IV), and on the molecular profile, and particularly on the presence of IDH (Isocitrate dehydrogenase) mutation which is associated with a better prognosis. Mutations of IDH1R132, less frequently IDH2R172 affect 40% of gliomas, mostly grade II and grade III. IDH mutation results in the accumulation of D-2 hydroxyglutarate (D2HG) produced by the IDH1 mutant enzyme. D2HG acts as a competitive inhibitor of the alphaketoglutarate cofactor in a wide range of cellular reactions, including TET family enzymes and histone demethylases, resulting in DNA hypermethylation (CpG Island Methylator Phenotype, CIMP) and histone hypermethylation. IDH mutation is probably the earliest genetic alteration in the tumorigenesis of gliomas, and is also the most stable, as shown in a whole exome analysis of initial and recurring low grade gliomas. It is therefore an attractive target. In an attempt to reverse the CIMP status, in vitro and in vivo experiments showed a dramatic anti-tumor effect of hypomethylating drugs (5-azacytidine and 5-deoxyazacytidine) on IDH1 mutated human gliomas . These hypomethylating drugs are routinely used in myelodysplasic syndrome and are well tolerated. Despite glioma with IDH1/2 mutation have a better outcome compared to the IDH wild-type counterpart, the prognosis remains grim with no therapeutic perspective after radiotherapy, temozolomide and/or nitrosourea treatment. Another reason to administer the hypomethylating drug after failure of alkylating chemotherapy is based on the assumption that demethylation of O6-methylguanine-DNA-methyltransferase (MGMT) promoter could compromise the efficacy of future alkylating treatment. Based on preclinical data obtained in animal models and clinical data of patients with MDS, we will treat with demethylating drug (Azacitidine, Vidaza®) patients with recurrent IDH mutated gliomas (as authentificated by IDHR132H Immunochemistry or direct sequencing). Preclinical data on experimental gliomas and clinical data on MDS, has shown that efficacy is delayed by three or more cycles. This has important consequences in the selection of the population, and the follow-up of the treatment. We will exclude patients with important mass effect and intracranial hypertension, and more generally patients whose life expectancy is inferior to 9 months. Despite such treatment has never been evaluated in IDH mutated glioma patients, the biological and preclinical backgrounds are extremely strong and the drug is well tolerated and widely used in the field of haematology.

Azacitidine is believed to exert its antineoplastic effects by multiple mechanisms including cytotoxicity on abnormal haematopoietic cells in the bone marrow and hypomethylation of DNA. The cytotoxic effects of azacitidine may result from multiple mechanisms, including inhibition of DNA, RNA and protein synthesis, incorporation into RNA and DNA, and activation of DNA damage pathways. Non-proliferating cells are relatively insensitive to azacitidine. Incorporation of azacytidine into DNA results in the inactivation of DNA methyltransferases, leading to hypomethylation of DNA.

DNA hypomethylation of aberrantly methylated genes involved in normal cell cycle regulation, differentiation and death pathways may result in gene re-expression and restoration of cancer suppressing functions to cancer cells. The relative importance of DNA hypomethylation versus cytotoxicity or other activities of azacitidine to clinical outcomes has not been established.

Azacitidine is small molecule. Pharmacokinetic data suggest a good penetration in the Central Nervous System (CNS). 5-aza-dCyd, active metabolite of azacitidine, can cross the blood-Cerebro Spinal Fluid (CSF) barrier effectively, producing cytotoxic concentrations in the CSF when given by i.v. infusion in animal models .

In IDH mutated tumors, it is believed that the inactivation of tumor suppressor genes by aberrant DNA methylation of CpG islands plays an important role in the development of malignancy. DNA methylation usually occurs at the 5-position of the cytosine ring within cytosine-phosphate-guanine (CpG) dinucleotide by a transfer of the methyl group from S-adenosyl-L-methionine. Azacitidine reactivates many tumor suppressor genes that are aberrantly silenced in hypermethylated tumors, including Rb, p53, CDKN2A, and mismatch repair genes which are involved in alkylating resistance. It may also reactivate MGMT, which makes the cell more sensitive to alkylating drugs: this may be a deleterious effect. This is one more reason to reserve this treatment to patients previously treated with alkylating drugs which developed secondary resistance: one of the mechanisms of resistance is the inactivation of mismatch repair genes which occurs after alkylating treatment and is a mechanism of secondary resistance in MGMT promoter methylated gliomas. Re-expressing these genes may render the tumor more sensitive to chemotherapy.

Description and justification of the dosage, route of administration, administration schedule and treatment duration:

Vidaza® is approved by the European Commission for the treatment of adult patients who are not eligible for haematopoietic stem cell transplantation (HSCT) with: intermediate-2 and high-risk myelodysplastic syndromes (MDS) according to the International Prognostic Scoring System (IPSS),, chronic myelomonocytic leukaemia (CMML) with 10-29 % marrow blasts without myeloproliferative disorder, acute myeloid leukaemia (AML) with 20-30 % blasts and multi-lineage dysplasia, according to World Health Organization (WHO) classification, AML with >30% marrow blasts according to the WHO classification.

In these approved indications, the recommended starting dose for the first treatment cycle, for all patients regardless of baseline haematology laboratory values, is 75 mg/m2 of body surface area, injected subcutaneously, daily for 7 days, followed by a rest period of 21 days (28-day treatment cycle) every 4 weeks until progression, intolerance or end of the study. It is recommended that patients be treated for a minimum of 6 cycles. In absence of study in neuro-oncology, it was decided to use same dosage and schedule as in haematological malignancies.

Summary of the known and foreseeable benefits and risks for the study participants:

In this population, there is currently no available treatment, shown to have any efficacy. Despite there is no data on efficacy of azacitidine in this population there is a strong biological and preclinical background. Furthermore the tolerance is well known since the drug is widely used in hematology. The toxicity is mostly haematologic and renal and easily manageable. However there are two caveats:

* Since the response is delayed, we expect no effect before 3 cycles. Moreover neurological worsening must be expected and anticipated and treated if necessary by introducing or increasing steroids.
* Demethylation modifies gene expression and reactivates tumor suppressor genes; however we cannot not exclude a deleterious effect (ie reactivation of deleterious genes). This is a theoretical risk though it has not been reported in the MDS and AML treated with azacitidine.

Objectives and endpoints:

The primary objective of this study will be to evaluate the efficacy based on RANO criteria, of azacitidine in patients with recurrent IDH1/2 mutated glioma after conventional treatments. The primary assessment criterion will be Progression-Free Survival at 6 months (PFS-6) (24 weeks) estimated by the RANO criteria.

The Secondary objectives will be 1/ to evaluate the clinical efficacy: objective response rate after 6 cycles of treatment evaluated by RANO criteria and overall survival, 2/ to evaluate the safety and tolerability of azacitidine by description and graduation of adverse events according to the revised NCI Common Terminology Criteria for Adverse Events (CTCAE V4.0).

Design of the Study:

The AGIR Trial will be a phase II, non-comparative, open label, non randomised monocentric trial evaluating efficacy of a treatment by azacitidine in recurrent IDH1/2 mutant gliomas.

Statistical aspects:

A Fleming two-stage design is used to assess the efficacy of Azacitidine on the 6-months progression free survival. Minimal efficacy (p0) and expected efficacy (p1) are respectively fixed to 15% and 30%. With a type I error rate of 5%, and an 80% power, 19 patients are required for the first step, and 36 additional patients for the second step if no conclusion has been reached at intermediate analysis. In this configuration we plan to enroll 63 patients in order to have 55 patients who will receive at least 1 cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Glioma grade II or III with IDH1 or IDH2 mutation
* Recurring after standard treatment, ie radiotherapy and at least one alkylating chemotherapy, or alkylating chemotherapy alone in case of gliomatosis cerebri
* For the patients treated by radiotherapy, recurrence occurring more than three months from the end of the radiotherapy or occurring outside the irradiated volume
* Karnofsky Performance Status > 50
* Life expectancy > 9 months
* Suitable laboratory values obtained ≤ 7 days before inclusion visit:

  * Absolute neutrophil count (ANC) ≥ 1500 /mm3
  * Leucocytes ≥ 3,0 x 109/L
  * Platelet count ≥ 75 000 / mm3
  * Hemoglobin > 9.0 g/dL
  * Serum GlutamoOxaloacetate Transferase (SGOT) (AST) ≤ 3 x Upper Limit of Normal (ULN)
  * Serum Glutamate Pyruvate Transaminase (SGPT) (ALT) ≤ 3 x ULN
  * Creatininemia ≤ 1.5 x ULN
  * Bicarbonates ≥ 22 mmol/l
* Women of child-bearing potential (i.e. women who are pre-menopausal or not surgically sterile) must :

  * Have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study.
  * Agree to use, and to be able to comply with, effective contraception without interruption, throughout the entire duration study drug therapy (including doses interruptions) and for 3 months after the end of the study drug therapy.
* Male patients :

  * must agree to use a condom if engaged in sexual activity with a woman of childbearing potential during the entire period of treatment and during 3 months after end of treatment.
  * are informed about the procedures for preservation of sperm before starting treatment.
* Written informed consent dated and signed, prior to any study specific procedures (sampling, treatment and analyses).
* Affiliation to the French health insurance (recipient or assign)

Exclusion Criteria:

* Breast-feeding women
* Any evidence of severe or uncontrolled systemic diseases (as judged by the investigator), including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV) (Screening for chronic conditions is not required)
* Active pulmonary disease or congestive cardiac insufficiency
* Malignant hepatic tumor at a later stage
* Intracranial hypertension or important deviation of the midline on the MRI
* Any investigational agents or study drugs from a previous clinical study (within 30 days before the first dose of study treatment
* Any chemotherapy, anticancer immunotherapy or anticancer agents within 4 weeks (6 weeks for nitrosourea) before the first dose of study treatment
* Any unresolved toxicities (excepted alopecia and lymphopenia), from prior therapy greater than CTCAE grade 1 at the time of inclusion
* Known hypersensitivity to Azacitidine or Mannitol (E421), (refer to the Investigator's Brochure)
* Patients under curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2024-03-23 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival at 6 months (PFS-6) | at Month 6 after first administration of the drug
  Evaluation of the efficacy based on Radiologic Assessment in Neuro-Oncology (RANO) criteria,

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | During all the study until 1 Month after the last administration of the drug
  Incidence of each adverse events and serious adverse events and graduation according to the revised NCI Common Terminology Criteria for Adverse Events (CTCAE V4.0).
Overall Response rate at 6 months | At the end of Cycle 6 (each cycle is 28 days)
  Objective response rate (partial response (PR) and complete response (CR) to total treatment duration for 6 months, or until progressive disease, unacceptable toxicity or withdrawal of consent.
Overall survival (OS) | Through study completion up to 42 months
  OS is defined as the number of days from the date of the first dose of azacitidine to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEHAIS, MD, Principal Investigator — Hospital Pitié-Salpêtrière, Paris
Locations (1):
- Pitie Salpetriere Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.